CLINICAL TRIAL: NCT04380259
Title: Mindfulness-Based Trauma Recovery for Refugees (MBTR-R): Efficacy, Safety and Mechanisms
Brief Title: Mindfulness-Based Trauma Recovery for Refugees (MBTR-R)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBTR-R Tel Aviv
Record Dates: First submitted 2020-04-26; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-04

CONDITIONS: Stress Disorders, Post-Traumatic; Stress Related Disorder
Keywords: Asylum Seekers, Anxiety, Compassion, Depression, Mindfulness, PTSD, Post-Migration Stress, Refugees, Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBTR-R (Mindfulness-Based Trauma Recovery for Refugees) (Experimental): Mindfulness-based group intervention consisting of nine 2.5-hour weekly sessions.
  Interventions: Behavioral: Mindfulness-Based Trauma Recovery for Refugees (MBTR-R)
- Waitlist-Control (No Intervention): Following the 9-week waitlist period and 1-week post-intervention assessment, participants randomized to waitlist-control were offered an equivalent group intervention (i.e., 22.5 total hours, group instructor and cultural mediator, psychoeducation and low-intensity cognitive behavior therapy skill training, relaxation techniques).

INTERVENTIONS:
Behavioral: Mindfulness-Based Trauma Recovery for Refugees (MBTR-R) — MBTR-R is a mindfulness-based group intervention of nine 2.5-hour weekly sessions. MBTR-R format and structure parallel MBSR (mindfulness-based stress reduction) and MBCT (mindfulness-based cognitive therapy). MBTR-R includes systematic training in formal and informal mindfulness practices with trauma-sensitive adaptations and home practice. Trauma-sensitive adaptations include a "safe place" practice, psychoeducation about posttraumatic stress, stress reactivity, as well as self-compassion practices to cope with fear, self-judgement, guilt and shame. Socio-cultural adaptations include real-time linguistic translation of each session by a cultural mediator from the refugee community and use of socio-culturally specific metaphors. MBTR-R groups were conducted for men and women separately and delivered in an accessible, "safe space" in the local refugee community. Group meetings included a shared meal of traditional Eritrean food and female participants were offered free child care.
  Arms: MBTR-R (Mindfulness-Based Trauma Recovery for Refugees)

SUMMARY:
Worldwide, refugees and asylum seekers suffer at high rates from trauma- and stress-related mental health problems. The investigators thus developed Mindfulness-Based Trauma Recovery for Refugees (MBTR-R) - a 9-week, mindfulness- and compassion-based, trauma-sensitive and socio-culturally adapted, group intervention for refugees and asylum seekers. The overarching aims of the study were to, first, test whether MBTR-R is an efficacious and safe mental health intervention for traumatized refugees and asylum seekers with respect to stress- and trauma-related mental health outcomes; and, second, to test theorized mechanisms of action of MBTR-R. Accordingly, the investigators conducted a randomized waitlist-controlled trial among a community sample of female and male Eritrean asylum seekers in an urban post-displacement setting in the Middle East (Israel).

DETAILED DESCRIPTION:
Broadly, the investigators aimed to assess whether MBTR-R is an efficacious and safe mental health intervention for traumatized asylum seekers. Aim I: The investigators predicted that, relative to a waitlist control condition, MBTR-R will lead to improved stress-and trauma-related mental health outcomes, including lower levels and rates of posttraumatic stress, depression, anxiety, and improved subjective well-being at post-intervention and 5-week follow-up. Aim II: The investigators aimed to test, whether relative to the waitlist-control condition, MBTR-R was safe and thus not associated with participant-level clinically significant deterioration in any of the monitored primary mental health outcomes at post-intervention or at follow-up. In the event of adverse responding, the investigators planned to test whether key demographic factors or pre-existing vulnerability factors at pre-intervention that may predict participant-level deterioration or adverse responding to the intervention - so as to identify candidate contraindications for MBTR-R. Aim III: The investigators predicted that, relative to a waitlist control condition, MBTR-R will lead to changes in psycho-behavioral processes targeted by the intervention and implicated in vulnerability at pre-intervention, from pre-to-post intervention, measured in controlled behavioral and cognitive-experimental lab tasks or experience sampling measures, including measures of (a) self-compassion and self-criticism, (b) self-referential processing of fear, (c) avoidance, (d) emotional reactivity to trauma-related information and autobiographical memory, (e) impaired executive functions of trauma-related information processing in working memory. Aim IV: The investigators aimed to test whether, among the MBTR-R group, pre-to-post-intervention change and pre-intervention to follow-up change in mental health outcomes (Aim I) will be predicted or mediated by pre-to-post intervention change in the targeted psycho-behavioral processes.

ELIGIBILITY:
Inclusion Criteria:

* Eritrean refugee or asylum seeker living in Israel

Exclusion Criteria:

* active suicidality
* current psychotic symptoms
* current mental health treatment (e.g. psychotherapy, participation in psycho-social support group)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-05-18 (Actual); Study Completion 2019-05-18 (Actual)

PRIMARY OUTCOMES:
Harvard Trauma Questionnaire (HTQ) | Change from 1-week pre-intervention to 1-week post-intervention and change from 1-week pre-intervention to 5-weeks post-intervention
  The Harvard Trauma Questionnaire (HTQ) is a 16-item self-report questionnaire to assess post-traumatic stress symptom severity (5-point Likert scale) with higher scores indicating greater post-traumatic stress severity (minimum scale score 1 and maximum scale score 5), HTQ mean cut-off score ≥ 2 is commonly used to identify categorical (diagnostic) symptom status of post-traumatic stress disorder
Brief Patient Health Questionnaire (PHQ-9) | Change from 1-week pre-intervention to 1-week post-intervention and change from 1-week pre-intervention to 5-weeks post-intervention
  The brief Patient Health Questionnaire (PHQ-9) is a 9-item self-report questionnaire to assess depression symptom severity (5-point Likert scale) with higher scores indicating greater depression symptom severity (minimum scale score 0 and maximum scale score 36), PHQ-9 mean cut-off score ≥10 is commonly used to identify categorical (diagnostic) symptom status of depression
Beck's Anxiety Inventory (BAI) | Change from 1-week pre-intervention to 1-week post-intervention and change from 1-week pre-intervention to 5-weeks post-intervention
  The Beck's Anxiety Inventory (BAI) is a 21-item self-report questionnaire to assess anxiety symptom severity (4-point Likert scale) with higher scores indicating greater anxiety symptom severity (minimum scale score 0 and maximum scale score 63), BAI total cut-off score ≥ 16 is commonly used to identify categorical (diagnostic) symptom status of anxiety disorder

SECONDARY OUTCOMES:
Brief Inventory of Thriving (BIT) | 1-week pre-intervention, 1-week post-intervention and 5-weeks post-intervention
  One item of the 9-item self-report questionnaire Brief Inventory of Thriving (BIT) was used to assess subjective well-being (5-point Likert scale) with higher scores indicating greater subjective well-being (minimum score 1 and maximum score 5)
Post-Migration Living Difficulties Checklist (PMLD) | 1-week pre-intervention
  The Post-Migration-Living-Difficulties Checklist (PMLD) is a 9-item self-report questionnaire to assess post-migration stress (5-point Likert scale) with higher scores indicating greater post-migration stress (minimum scale score 1 and maximum scale score 5)
The State Shame and Guilt Scale (SSGS) | 1-week pre-intervention, 1-week post-intervention and 5-weeks post-intervention
  The State Shame and Guilt Scale (SSGS) is a 15-item self-report questionnaire to assess state shame and guilt (5-point Likert scale) with higher scores indicating greater levels of state shame, guilt and pride (minimum scale score 15 and maximum scale score 75)
The Short Self Compassion Scale (SSCS) | 1-week pre-intervention, 1-week post-intervention and 5-weeks post-intervention
  The Short Self-Compassion Scale SSCS is a 12-item self-report questionnaire to assess different facets of self-compassion (5-point Likert scale) with higher scores indicating greater levels of self-compassion (minimum scale score 1 and maximum scale score 5)
The Five Facets Mindfulness Questionnaire (FFMQ) | 1-week pre-intervention, 1-week post-intervention and 5-weeks post-intervention
  The Five Facets of Mindfulness Questionnaire (FFMQ) is a self-report questionnaire to assess different facets of trait mindfulness (5-point Likert scale) with higher scores indicating greater levels of trait mindfulness (minimum scale score 1 and maximum scale score 5)
Moral Injury Event Scale | 1-week pre-intervention, 1-week post-intervention and 5-weeks post-intervention
  The Moral Injury Event Scale is a self-report questionnaire to assess moral injury (6-point Likert scale) with higher scores indicating greater levels of moral injury (minimum scale score 1 and maximum scale score 6)
Trauma Cue Exposure Task | 1-week pre-intervention, 1-week post-intervention
  The Trauma Cue Exposure Task measures behavioral avoidance in response to trauma cues
Autobiographical Memory Recall Task | 1-week pre-intervention, 1-week post-intervention
  The Autobiographical Memory Recall Task measures avoidance in response to recalling a traumatic autobiographical memory
Adapted Sternberg Working Memory Task | 1-week pre-intervention, 1-week post-intervention
  The Adapted Sternberg Working Memory Task measures working memory processing of trauma- and stress-related words versus positive words
Self-Referential Encoding Task (SRET) of Self-Compassion and Self-Criticism | 1-week pre-intervention, 1-week post-intervention
  The SRET measures self-referential processing of self-criticism and self-compassion
Single Experience and Self-Implicit Association Task (SES-IAT) | 1-week pre-intervention, 1-week post-intervention
  The SES-IAT measures self-referential processing of fear
Experience Sampling of State Mindfulness | 15-minutes pre-intervention session and 15-minutes post-intervention session
  3-item experience sample (5-point Likert scale) of state mindfulness (minimum score 3 maximum score 15), higher scores indicate greater levels of state mindfulness
Experience Sampling of Cognitive Avoidance | 15-minutes pre-intervention session
  1-item experience sample (5-point Likert scale) of cognitive avoidance (minimum score 1 maximum score 5), higher scores indicate greater levels of cognitive avoidance
Experience Sampling of Negative Repetitive Thinking | 15-minutes pre-intervention session
  1-item experience sample (5-point Likert scale) of negative repetitive thinking (minimum score 1 maximum score 5), higher scores indicate greater levels of negative repetitive thinking
Experience Sampling of Emotion | 15-minutes pre-intervention session and 15-minutes post-intervention session
  4-item experience sample (5-point Likert scale) of the emotions happy, calm, sad and nervous/tense (minimum score 4 maximum score 20), higher scores indicate greater levels of the emotions happy, calm, sad and nervous/tense
Experience Sampling of Formal and Informal Mindfulness Practice | 15-minutes pre-intervention session
  2-item experience sample number of formal and informal mindfulness practice during the past week, higher scores indicate greater number of mindfulness practices during the past week
Experience Sampling of Self-Compassion | 15-minutes pre-intervention session
  1-item experience sample (5-point Likert scale) of negative self-compassion (minimum score 1 maximum score 5), higher scores indicate greater levels of self-compassion
Experience Sampling of Depression | 15-minutes pre-intervention session
  1-item experience sample (5-point Likert scale) of depression (minimum score 1 maximum score 5), higher scores indicate greater levels of depression
Experience Sampling of Anxiety | 15-minutes pre-intervention session
  1-item experience sample (5-point Likert scale) of anxiety (minimum score 1 maximum score 5), higher scores indicate greater levels of anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Amit Bernstein, Principal Investigator — University of Haifa
Locations (1):
- Kuchinate, Tel Aviv, Central District, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oren-Schwartz R, Aizik-Reebs A, Yuval K, Hadash Y, Bernstein A. Effect of mindfulness-based trauma recovery for refugees on shame and guilt in trauma recovery among African asylum-seekers. Emotion. 2023 Apr;23(3):622-632. doi: 10.1037/emo0001126. Epub 2022 Aug 4. PMID 35925708
- [Derived] Blay Benzaken Y, Zohar S, Yuval K, Aizik-Reebs A, Gebremariam SG, Bernstein A. COVID-19 and Mental Health Among People Who Are Forcibly Displaced: The Role of Socioeconomic Insecurity. Psychiatr Serv. 2023 Feb 1;74(2):158-165. doi: 10.1176/appi.ps.202200052. Epub 2022 Jul 14. PMID 35833254
- [Derived] Aizik-Reebs A, Amir I, Yuval K, Hadash Y, Bernstein A. Candidate mechanisms of action of mindfulness-based trauma recovery for refugees (MBTR-R): Self-compassion and self-criticism. J Consult Clin Psychol. 2022 Feb;90(2):107-122. doi: 10.1037/ccp0000716. PMID 35343723